CLINICAL TRIAL: NCT02286271
Title: Preliminary Testing of a Novel Device to Detect Epileptic Seizures
Acronym: PTEpD
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIP version 5.1
Record Dates: First submitted 2014-11-04; First posted 2014-11-07 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2016-08

CONDITIONS: Epilepsy
Keywords: Seizure detection
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Official statistics report around 1000 deaths due to epilepsy in the UK each year (Hanna et al 2002). Most of these deaths are un-witnessed and in many cases are believed to have been avoidable with timely assistance (Langan et al 2000). A major problem is detecting nocturnal seizures to allow body re-positioning, to maintain an open airway and to administer rescue medication. There are several seizure alarms commercially available but are often unreliable with many false alarms. The aim of this study is to investigate a novel seizure detection system with a unique algorithm.

DETAILED DESCRIPTION:
Two duplicate novel medical devices conforming to safety regulation BS EN 60601 containing the unique algorithm will be evaluated in clinical trials at two hospitals over a 14 month period. Each device is time synchronised with an Electroencephalographic (EEG) videotelemetry system which is the gold standard in identifying different seizure types recording from scalp electrodes. The devices will be monitoring participants from 3 months and older (children and adults). The algorithm was created from results from a PhD where 527 seizures were categorised into different seizure types. Sensitivity of identifying seizures was 91% and specificity was 75% using an optimal trigger level and algorithm. This trial will investigate how reliable the algorithm is in practice and determine an optimal trigger level..

ELIGIBILITY:
Inclusion Criteria:

* Frequent epileptic seizures 3 months and older Informed consent for participation

Exclusion Criteria:

* Infrequent seizures Attacks are of a non-epileptic nature Younger than 3 months Has an implantable device No informed consent.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are being admitted for electroencephalographic videotelemetry as part of their clinical management of their epilepsy will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Reliable detection of epileptic seizures (Trigger level to be determined for total seizures) | 14 months
  Trigger level to be determined for total seizures

SECONDARY OUTCOMES:
Reliable detection of epileptic seizures (Trigger level to be determined for different types of seizures.) | 14 months
  Trigger level to be determined for different types of seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Peter AG Sandercock, BA,BM, BCh, Study Chair — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Western General Hospital, Edinburgh
  - Royal Hospital for Sick Children, Edinburgh

REFERENCES:
- [Background] Hanna H.J, Black M, Sander J.W.S, Smithson W.H, Appleton R, Brown S, Fish D.R. The National Sentinel Clinical Audit of Epilepsy-Related Death- Death in the Shadows. The Stationery Office. The National Sentinel of Epilepsy-Related Deaths Report 2002 ISBN 0-117-02868-1
- [Background] Langan Y, Nashef L, Sander JW. Sudden unexpected death in epilepsy: a series of witnessed deaths. J Neurol Neurosurg Psychiatry. 2000 Feb;68(2):211-3. doi: 10.1136/jnnp.68.2.211. PMID 10644790